CLINICAL TRIAL: NCT07066826
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Placebo- and Active-Controlled, Parallel-Group Phase II/III Clinical Study to Evaluate the Efficacy and Safety of Huperzine A Controlled-Release Tablets in Patients With Mild-to-Moderate Dementia of the Alzheimer's Type
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Huperzine A Controlled-Release Tablets in Patients With Mild-to-Moderate Dementia of the Alzheimer's Type
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wanbangde Pharmaceutical Group Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WanbangdePharm1
Record Dates: First submitted 2025-07-01; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Dementia
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Huperzine A controlled-release tablets (Experimental)
  Interventions: Drug: Huperzine A Controlled-Release Tablets
- Donepezil hydrochloride tablets (Active Comparator)
  Interventions: Drug: Donepezil hydrochloride tablets
- Huperzine A controlled-release tablets placebo; Donepezil hydrochloride tablets placebo (Placebo Comparator)
  Interventions: Drug: Huperzine A controlled-release tablets placebo; Donepezil hydrochloride tablets placebo

INTERVENTIONS:
Drug: Huperzine A Controlled-Release Tablets — During the trial, the patients should take huperzine A controlled-release tablets in the morning
  Arms: Huperzine A controlled-release tablets
Drug: Donepezil hydrochloride tablets — During the trial, the patients should take donepezil hydrochloride tablets before going to bed in the evening
  Arms: Donepezil hydrochloride tablets
Drug: Huperzine A controlled-release tablets placebo; Donepezil hydrochloride tablets placebo — During the trial, the patients should take huperzine A controlled-release tablets placebo in the morning and donepezil hydrochloride tablets placebo before going to bed in the evening
  Arms: Huperzine A controlled-release tablets placebo; Donepezil hydrochloride tablets placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, double-dummy, active- and placebo-controlled, parallel-group clinical trial. The dose confirmation stage is designed to evaluate the efficacy and safety of different doses of huperzine A controlled-release tablets in patients with mild-to-moderate dementia of the Alzheimer's type, with the goal of providing a basis for dose selection in the subsequent efficacy confirmation stage. The efficacy confirmation stage aims to assess the effect of huperzine A controlled-release tablets on cognitive function and functional abilities in patients with mild-to-moderate dementia of the Alzheimer's type.In the open-label extension stage, all subjects will receive huperzine A controlled-release tablets until Week 52, to further evaluate the long-term efficacy and safety of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily agrees to participate in the study and signs the informed consent form jointly with a legally authorized representative (LAR). If the subject is unable to sign due to cognitive impairment or other reasons, the signature field for the subject may be left blank, with the reason specified and signed by the LAR. In such cases, the LAR must sign the informed consent form on behalf of the subject.
2. Aged ≥50 and ≤85 years, male or female.
3. Meets the diagnostic criteria for probable Alzheimer's disease (AD) dementia according to the 2011 National Institute on Aging and Alzheimer's Association (NIA-AA) guidelines.
4. Has experienced memory impairment for at least 12 months, with a chronic and progressively worsening course.
5. Has received ≥5 years of formal education and is able to complete the protocol-specified cognitive assessments.
6. Diagnosed with Stage 4 or 5 (mild to moderate dementia) according to the Revised Clinical Staging of Alzheimer's Disease (2024) (i.e., Clinical Dementia Rating [CDR] global score of 1 or 2).
7. Total score on the Mini-Mental State Examination (MMSE) is between 11 and 26 inclusive.
8. Has undergone a cranial MRI scan showing a Medial Temporal Atrophy (MTA) visual rating scale grade ≥1. If the subject has completed an eligible MRI at this or another tertiary hospital within 6 months prior to screening, and it meets the protocol requirements, re-scanning is not required.
9. Capable of undergoing positron emission tomography (PET) imaging.
10. Hachinski Ischemic Score (HIS) ≤ 4.
11. Hamilton Depression Rating Scale (HAMD-17) score of ≤10.
12. No obvious focal neurological signs on physical examination, except those attributable to peripheral injury.
13. Has a stable and reliable caregiver, or is in frequent contact with a caregiver (at least 4 days per week and ≥2 hours per day). The caregiver must accompany the subject to study visits, provide reliable information for scale assessments based on sufficient interaction and communication with the subject, and should remain the same throughout the study whenever possible.

Exclusion Criteria:

1. Subjects who are allergic to the active ingredient or excipients of huperzine A controlled-release tablets or donepezil, or those with lactose intolerance.
2. Cognitive impairment or dementia not caused by Alzheimer's disease (AD), including:

(1) Other neurodegenerative diseases (e.g., dementia with Lewy bodies, frontotemporal degeneration, Huntington's disease, Parkinson's disease); (2) Non-degenerative neurological conditions causing cognitive impairment or dementia (e.g., vascular cognitive impairment or dementia, hydrocephalus, encephalitis, hypoxic brain injury, traumatic brain injury); (3) Non-neurological systemic diseases causing cognitive impairment or dementia (e.g., endocrine disorders such as hypothyroidism, hepatic insufficiency, hepatic encephalopathy, dialysis encephalopathy, neurosyphilis, HIV); (4) Cognitive impairment or dementia caused by vitamin deficiencies (e.g., folate or vitamin B12 deficiency).

3.Subjects diagnosed, per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), with psychiatric disorders within the past 12 months that are unstable or may interfere with study assessments, including but not limited to schizophrenia or other psychotic disorders, bipolar disorder, major depressive disorder, delirium, or substance (including alcohol) use disorders with dependence.

4.Subjects with significant focal brain lesions on MRI, including but not limited to any of the following (if a qualifying head MRI was performed within 6 months prior to screening and meets protocol requirements, repeat imaging is not required):

1. Presence of lesions indicating large-area cerebral infarction;
2. Infarcts in critical brain regions (e.g., thalamus, hippocampus, entorhinal cortex, parahippocampal gyrus, angular gyrus, cortical or subcortical gray matter nuclei);
3. More than two infarcts with a diameter >2 cm, and deemed by the investigator to impact cognitive assessments;
4. Multiple lacunar infarcts, deemed by the investigator to impact cognitive assessments;
5. Severe white matter lesions;
6. Intracerebral hemorrhage deemed likely to affect cognitive assessments by the investigator;
7. Hydrocephalus.

5.Subjects with uncontrolled seizures (and/or epilepsy syndromes), or those with cognitive impairment caused or potentially caused by recurrent seizures or antiepileptic drug use.

6.Subjects who experienced acute cardiovascular or cerebrovascular events within 3 months prior to screening (e.g., unstable angina, second- or third-degree atrioventricular block or other serious arrhythmias, myocardial infarction, decompensated congestive heart failure of NYHA class III or IV, transient ischemic attack, or ischemic stroke).

7.Subjects with uncontrolled hypertension or hypotension at screening (defined as systolic blood pressure ≥160 mmHg or <90 mmHg, or diastolic blood pressure ≥100 mmHg or <60 mmHg after pharmacologic or non-pharmacologic treatment); subjects with slight deviations beyond this range but deemed clinically insignificant by the investigator may be included.

8.Subjects with serious active gastrointestinal disorders (e.g., severe gastroesophageal reflux, gastrointestinal bleeding, or peptic ulcers) within 3 months prior to screening, or who have undergone any surgical procedures that may affect drug absorption (e.g., total gastrectomy, total small bowel resection).

9.Subjects with other uncontrolled clinical conditions (e.g., malignancies, severe infectious diseases, respiratory diseases).

10.Subjects with sinus bradycardia at screening (resting heart rate <60 bpm) that is deemed clinically significant by the investigator.

11.Subjects with corrected QT interval using Fridericia's formula (QTcF) >450 ms in males or >470 ms in females at screening or baseline.

12.Subjects with renal dysfunction (serum creatinine [Scr] >1.5× the upper limit of normal [ULN] per the study center laboratory) or hepatic dysfunction (ALT or AST >2× ULN).

13.Subjects with thyroid function abnormalities at screening that are deemed clinically significant and unsuitable for study participation by the investigator.

14.Subjects who test positive for syphilis antibodies or HIV antibodies. 15.Subjects who received donanemab within 2 months prior to screening; lecanemab within 5 weeks prior to screening; or any other medication for the treatment of AD or cognitive enhancement within 4 weeks prior to screening, including but not limited to cholinesterase inhibitors, NMDA receptor antagonists, and other nootropic agents.

16.Subjects who participated in any drug clinical trial (excluding vitamins and minerals) within 1 month prior to screening or 7 half-lives of the study drug (whichever is longer), or who are currently participating in another clinical trial.

17.Subjects who are unable to complete the required scale assessments due to uncorrectable vision or hearing impairments.

18.Subjects who are unable to complete study-required assessments due to personal limitations, such as contraindications to MRI scanning.

19.Subjects of childbearing potential (male or female) who are unwilling to use effective contraception from the start of the study until 6 months after the end of the study, and/or female subjects of childbearing potential who are unwilling or unable to undergo pregnancy testing.

20.Pregnant or breastfeeding women. 21.Any other condition that, in the opinion of the investigator, renders the subject unsuitable for participation in the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-08-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
ADAS-Cog11 | week24
  ADAS-Cog11: Alzheimer's Disease Assessment Scale-Cognitive Subscale. Score range: 0-70. Lower = better
ADCS-ADL | week24
  ADCS-ADL: Alzheimer's Disease Cooperative Study - Activities of Daily Living. Score range: 0-78. Higher= better